CLINICAL TRIAL: NCT01908465
Title: Peripheral Histamine 1 Receptor Blockade in IBS
Brief Title: Peripheral Histamine 1 Receptor Blockade in IBS: Multicenter Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Guy Boeckxstaens, Prof. Dr., KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S55485
Record Dates: First submitted 2013-07-19; First posted 2013-07-25 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Irritable Bowel Syndrome (IBS)
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — ebastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ebastine (Active Comparator): Ebastine
  Interventions: Drug: Ebastine
- placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ebastine
  Arms: Ebastine
Drug: Placebo
  Arms: placebo

SUMMARY:
Purpose:

To evaluate the efficiency of Irritable Bowel Syndrome (IBS) patients treatment with the H1-receptor antagonist ebastine.

Design:

Double blind randomized placebo controlled trial. IBS patients receive a 12-weeks treatment with ebastine 20mg once daily or placebo (1:1 randomization).

ELIGIBILITY:
Inclusion Criteria:

* Irritable Bowel Syndrome (IBS) (ROME III criteria): subtype with diarrhea or mixed form
* age 18-65 years

Exclusion Criteria:

* IBS subtype with constipation
* medication: antidepressants or H1-receptor antagonists
* pregnancy, breast feeding
* co-morbidity: severe kidney- and/or liver disease or other gastrointestinal diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-11; Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Effect of treatment on global symptom relief (of IBS complaints) | after 12 weeks treatment
  By mean of weekly GSRS (Gastrointestinal Symptom Rating Scale )questionnaires and weekly "SGA (Subject's Global Assessment) of relief" and "SGA of Abdominal Pain and Discomfort" questionnaires

SECONDARY OUTCOMES:
Effect of treatment on stool consistency and frequency and other common IBS associated complaints (flatulence, urgency,...) | fter 12 weeks treatment
  By mean of weekly questionnaires

OTHER OUTCOMES:
Effect of treatment on quality of life | after 12 weeks treatment
  By mean of 'Quality of life" questionnaire (completed at the end (after 14 weeks) and the start of the study and after 8 and 12 weeks of treatment)
Effect of treatment on inflammatory mediators/metabolites in urine | after 12 weeks
  By metabolic profiling in urine samples before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Guy Boeckxstaens, M.D., Principal Investigator — Catholic University Leuven and Universitary Hospitals Leuven
Locations (12):
- Belgium (6):
  - UZ Antwerpen, Edegem, Antwerpen
  - ZOL (Ziekenhuis Oost-Limburg), Genk, Limburg
  - UZ Gent, Ghent, Oost-Vlaanderen
  - AZ Sint-Elizabeth Zottegem, Zottegem, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams-Brabant
  - AZ Sint-Lucas Brugge, Bruges, West-Vlaanderen
- Netherlands (6):
  - Rijnstate, Arnhem, Gelderland
  - Medisch Spectrum Twente, Enschede, Limburg
  - AZ Maastricht, Maastricht, Limburg
  - Sint Lucas Andreas Ziekenhuis, Amsterdam, North Holland
  - Academisch Medisch Centrum, Amsterdam, North Holland
  - Tergooiziekenuizen Blaricum/Hilversum, Blaricum, North Holland

REFERENCES:
- [Derived] Decraecker L, De Looze D, Hirsch DP, De Schepper H, Arts J, Caenepeel P, Bredenoord AJ, Kolkman J, Bellens K, Van Beek K, Pia F, Peetermans W, Vanuytsel T, Denadai-Souza A, Belmans A, Boeckxstaens G. Treatment of non-constipated irritable bowel syndrome with the histamine 1 receptor antagonist ebastine: a randomised, double-blind, placebo-controlled trial. Gut. 2024 Feb 23;73(3):459-469. doi: 10.1136/gutjnl-2023-331634. PMID 38191268